CLINICAL TRIAL: NCT06167499
Title: Impact of Therapeutic Education Consultations Conducted by Specialized Nurses on Glycemic Control and Quality of Life in Diabetic Patients Treated With Intensified Insulin Therapy: a Randomized Study
Brief Title: Therapeutic Education Consultations With Diabetic Patients Treated With Intensified Insulin Therapy
Acronym: DIABETE COACH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-05-DIABETE COACH
Record Dates: First submitted 2023-11-24; First posted 2023-12-12 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Diabete Mellitus; Insulin Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic Education Group. (Experimental): Medical follow-up every 6 months for 18 months (inclusion, M6, M12, M18) associated with therapeutic education consultations conducted by nurses in the month following inclusion (between D0 and M1), M3, M9 and M15
  Interventions: Other: Diabetes Therapeutic Education conducted by nurses
- Standard (No Intervention): Medical follow-up every 6 months for 18 months (Inclusion, M6, M12, M18) :usual practice

INTERVENTIONS:
Other: Diabetes Therapeutic Education conducted by nurses — Individual consultations with the therapeutic education IDE, who will help the patient to achieve the therapeutic objectives set before the medical consultation.
  Once the objectives have been set, the IDE will set up individual workshops and subsequently assess the patient's learning and its impact on his or her care. These workshops can include equipment demonstrations and practical exercises, explanations of treatment adaptation protocols, and dietary or sexual advice.
  Arms: Therapeutic Education Group.

SUMMARY:
Diabetes is a chronic condition that affects around 8% of the French population, and is associated with severe complications. Maintaining a constant blood glucose level of between 0.7 and 1.80 g/l is the day-to-day objective of diabetic patients.Insulin can be administered by injection via syringes or pens, or by insulin pumps and patients can perform self-monitoring of blood glucose.

All these actions can be the subject of therapeutic education, which involves a range of tools, including dedicated individual consultations carried out by state-qualified nurses.

The aim of the study is to evaluate the benefit of therapeutic education consultations conducted by nurses in addition to medical consultations, on the follow-up of diabetic patients, insulin pump carriers or treated with multiple injections, in terms of glycemic control, quality of life and medical complications. The objective of the study is to evaluate whether the therapeutic education consultations conducted by nurses can improve the care of the diabetic patient.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man aged 18 to 75
* Diabetic patient type 1 or 2 insulin-dependent
* Patient treated with multi-injections or insulin pump
* Patient equipped with FreeStyle Libre flash glucose monitoring system
* Glycemic imbalance with HBA1c > 8
* Patient living at home

Exclusion Criteria:

* Recent discovery (< 6 months) of diabetes
* Major intellectual disability
* Social isolation
* IMC > 35
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Rate of glycated hemoglobin HBA1c | 12 months
  Difference in HBA1c between baseline and 12 months (M12)

SECONDARY OUTCOMES:
Evaluation of glycemic control over 18 months | 18 months
  Evaluation via Freestyle free blood glucose sensor with free view software every 6 months, over the last month and the last 3 months prior to medical consultation:
  * % of time spent in target range (0.7 g/l ≤ blood glucose ≤ 1.8g/l)
  * % of time spent in hypoglycemia (blood glucose <0.7 g/l,
  * % of time spent in hyperglycemia (blood glucose > 1.8g/l) Recording of ketoacidosis episodes during patient attendance Recording of episodes of severe hypoglycemia requiring third-party assistance with the patient HBA1c monitoring every 3 months
Evaluation of patients' quality of life over 18 months | 18 months
  Questionnaire assessing quality of life (Audit of Diabetes Dependent Quality of Life - 19 items: ADDQoL 19)
Evaluation of patients' satisfaction with diabetes treatment | 18 months
  Questionnaire assessing satisfaction with diabetes treatment (Diabetes Treatment Satisfaction Questionnaires: DTSQs)
Evaluation of long-term complications over 18 months | 18 months
  Assessment of the development and evolution of diabetes-related complications: neuropathy, nephropathy, retinopathy, arteriopathy, erectile dysfunction, heart disease, hypertension, foot ulcers, amputations and cerebrovascular damage.
  Number of additional hospitalizations and urgent consultations for acute or chronic complications.

CONTACTS AND LOCATIONS:
Overall Officials: Elena BOUCHEZ, Principal Investigator — Hopital Nord Franche-Comte
Locations (1):
- Hôpital Nord Franche-Comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: No